CLINICAL TRIAL: NCT05524051
Title: A Randomized, Multi-centric, Placebo-controlled, Participant and Investigator-blinded Study to Evaluate the Safety, Tolerability and Efficacy of TIN816 in Adult Patients at Risk for Acute Kidney Injury Following Cardiac Surgery.
Brief Title: A Multi-center Study to Evaluate the Safety, Tolerability and Efficacy of TIN816 in Patients at Risk for Acute Kidney Injury Following Cardiac Surgery.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTIN816A12201; 2024-511621-64-00 (Other: EU CT)
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Acute Kidney Injury Following Cardiac Surgery
Keywords: acute kidney injury; cardiac surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TIN816 (Experimental): TIN816
  Interventions: Drug: TIN816
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TIN816 — TIN816
  Arms: TIN816
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, multi-centric, placebo-controlled, participant and investigator-blinded study to evaluate the safety, tolerability and efficacy of TIN816 in adult patients at risk for acute kidney injury following cardiac surgery.

DETAILED DESCRIPTION:
This is a randomized, multi-centric, placebo-controlled, participant and investigator-blinded study to evaluate the safety, tolerability and efficacy of TIN816 in adult patients at risk for acute kidney injury following cardiac surgery. The screening period will last up to 30 days and the whole study will last up to 120 days. Approximately 120 subjects will be randomized to TIN816 or placebo. Efficacy will be evaluated 5 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Participants must be able to communicate well with the investigator and to understand and comply with the requirements of the study.
* Male and female patients ≥45 years at screening.
* Participants must weigh at least 50 kg and maximum 150 kg to participate in the study and must have a body mass index (BMI) below 40. BMI = Body weight (kg) / [Height (m)]2.
* At screening, vital signs should be assessed in the sitting or supine position and be within the following ranges:

  1. body temperature between 35.0-37.5 °C
  2. blood pressure (systolic 100-160 mmHg, diastolic < 100 mmHg)
  3. pulse rate (50-100/min) stable with or without medication(s) as per Investigator assessment.
* No known increase in SCr of ≥25% at screening visit compared to a previous value obtained within the last 6 months as documented by a local laboratory using standard assay methodology.
* Non-emergent open chest cavity major cardiopulmonary bypass (CPB) surgery with expected CPB time ≥1 hour

Exclusion Criteria:

* eGFR at screening <15 mL/min/1.73 m2 (calculated using CKD-EPI 2021 equation).
* Receiving renal replacement therapy currently or at any time within 3 months prior to screening.
* Patients with bleeding risk at screening. The Investigator should make this determination in consideration of the participant's medical history and/or clinical or laboratory evidence of any of the following:

  * History of bleeding with suspected or confirmed bleeding disorder or any other high risk for bleeding in the opinion of the investigator
  * Thrombocytopenia: platelet count< 100x109/L
  * History of platelet dysfunction: e.g., ADP induced platelet aggregation lower than 60 %
  * History of coagulation factor deficiency: including, but not limited to fibrinogen ≤ 2.5 g/L or Von Willebrand factor (vWF) ≤ 50 IU/dL
* Any emergency surgeries performed less than 30 days before screening, including aortic dissection, and/or major congenital heart defects.
* Scheduled to undergo cardiac surgery off CPB or with hypothermic circulatory arrest.
* Cardiogenic shock or hemodynamic instability within four weeks prior to surgery, requiring inotropes or vasopressors or mechanical devices such as intra-aortic balloon counter-pulsation (IABP).
* Have received cardiopulmonary resuscitation (CPR) within 30 days prior to cardiac surgery.
* Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or until the expected PD effect has returned to baseline, whichever is longer; or longer if required by local regulations.
* Patients who are post-nephrectomy
* Have ongoing sepsis or history of sepsis within the past 8 weeks or untreated diagnosed infection prior to screening visit. Sepsis is defined as presence of a confirmed pathogen, along with fever or hypothermia, and hypoperfusion or hypotension.
* Recent (within the last three years) and/or recurrent history of autonomic dysfunction (e.g., recurrent episodes of fainting, palpitations, etc.).
* Pregnant or nursing (lactating) women
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception while taking study treatment and until the end of study. Highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g. calendar, symptothermal and post-ovulation methods) and withdrawal are not acceptable methods of contraception.
  * Female bilateral tubal ligation, female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or total hysterectomy at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
  * Male sterilization (at least 6 months prior to screening). For female participants on the study, the vasectomized male partner should be the sole partner for that participant.
  * Use of oral (estrogen and progesterone), injected, or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception.

Ages: 45 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Ratio of the highest serum creatinine value up to and including Study Day 6 versus baseline | from baseline to Day 6
  To assess the effect of TIN816 on serum creatinine level in high-risk patients undergoing major cardio-vascular surgery, versus placebo

SECONDARY OUTCOMES:
AKI stages 1, 2 and 3 as defined by modified AKI Network criteria | from baseline to Day 6
  To assess the effect of TIN816 on the incidence and severity of AKI in patients at high risk for AKI and undergoing major cardio-vascular surgery, versus placebo
Anti-drug antibodies against TIN816 | from baseline to 90 Days
  To assess immunogenicity (IG) of TIN816
Occurrence of major adverse kidney event at Day 90 (MAKE90) | 90 Days
  To assess the effect of TIN816 on the incidence of AKD in high-risk patients undergoing major cardio-vascular surgery, versus placebo
Occurrence of MAKE30 | 30 Days
  To assess the effect of TIN816 on the incidence of AKD in high-risk patients undergoing major cardio-vascular surgery, versus placebo
Occurrence of individual components of the MAKE criteria at Days 30 or 90. | 30 or 90 Days
  To assess the effect of TIN816 on the incidence of AKD in high-risk patients undergoing major cardio-vascular surgery, versus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticasl
Locations (34):
- United States (2):
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - Duke Univ Medical Center, Durham, North Carolina
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, CABA
- Belgium (2):
  - Novartis Investigative Site, Genk, Limburg
  - Novartis Investigative Site, Leuven
- Brazil (2):
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Salvador
- Canada (2):
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Novartis Investigative Site, Ostrava, Poruba, Czechia
- Novartis Investigative Site, Tartu, Estonia
- France (5):
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Neuilly-sur-Seine
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Rennes
- Germany (4):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Essen
- Hungary (3):
  - Novartis Investigative Site, Pécs, Baranya
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Budapest
- India (2):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
- Novartis Investigative Site, Vilnius, Lithuania
- Novartis Investigative Site, Singapore, Singapore
- Spain (4):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Badalona, Barcelona
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com